## Avatar trial protocol -Amendment to surgical delays-

Aortic Valve Replacement Versus Conservative Treatment in Asymptomatic Severe Aortic Stenosis (AVATAR trial)

NCT number: NCT02436655.

Date of amendment: 04.01.2021

## Amendmen to statystical analysis

- 1. Patients randomized to AVR surgery who received delayed surgery (more than 8 weeks after randomization) due to COVID -19 public health emergency will be documented and this delay will be defined as an anticipated minor deviation from the clinical protocol
- 2. Appropriate statistical procedures will be performed and results will be published according to the FDA guidance "Conduct of Clinical Trials of Medical Products During the COVID-19 Public Health Emergency Guidance for Industry, investigators, and Institutional Review Boards"